CLINICAL TRIAL: NCT06370299
Title: Screening of Multidrug Resistant Bacteria, and the Implication of a Positive Screening Result Compared to a Negative on Subsequent Infection and Mortality.
Brief Title: Screening of Multidrug Resistant Bacteria, and the Clinical Implication for the Patient
Status: Not yet recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-06402-01
Record Dates: First submitted 2024-03-07; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-02

CONDITIONS: Multi-antibiotic Resistance
Keywords: Multidrug Resistance; Acinetobacter baumannii; Pseudomonas aeruginosa; carbapenem-resistant; gram-negative resistance; ESBL; carbapenemase-producing Enterobacterales; colonization; screening
MeSH Terms: conditions — Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients screened for MDR gram negative bacilli with positive detection: This group has risk factors for acquisition of multidrug resistant gram negative bacilli (e.g hospital admission outside of Scandinavia), and are therefore screened. They have a detection of ESBL producing Enterobacterales (EPE), Carbapenemase producing Enterobacterales (CPE), Carbapenem resistant A.baumannii (CRAB) and/or carbapenem resistant P.aeruginosa (CRPA).
  Interventions: Other: (exposure of) MDR carriage
- patients screened for MDR gram negative bacilli with negative detection: This group has also similar risk factors for acquisition of multidrug resistant gram negative bacilli (e.g hospital admission outside of Scandinavia), and are therefore screened, but they do not have a detection of EPE, CPE, CRAB and/or CRPA.

INTERVENTIONS:
Other: (exposure of) MDR carriage — The difference in exposure between the two groups is the carriage or non-carriage of multidrug resistant gram negative bacilli.
  Groups: patients screened for MDR gram negative bacilli with positive detection

SUMMARY:
The goal of this observational study is to evaluate the screening for multidrug resistant bacteria in patients admitted to hospitals in Scania. The main questions it aims to answer are:

* admission rates after screening
* 30-day and one-year mortality after screening Participants will be evaluated for positive screening results with following multidrug resistant gram negative bacilli: ESBL producing Enterobacterales, Carbapenemase producing Enterobacterales, Carbapenem resistant P.aeruginosa and carbapenem resistant Acinetobacter baumannii. Researchers will compare patients with positive and negative screening results to see, if the relative risks in the two groups differ in admission rates and mortality.

DETAILED DESCRIPTION:
Infections with multidrug resistant bacteria (MDR) cause more than one millions deaths globally according to World Health Organisation. While Scandinavia is still a low-endemic area of resistance compared to other parts of the world, such as South-Asia, South-Europe, a worrisome rise in MDR has been observed in the past decade. Of concern is particularly gram negative bacilli, e.g extended spectrum beta-lactamase (ESBL) and carbapenemase producing Enterobacterales (EPE and CPE) as well as carbapenem resistant Pseudomonas aeruginosa (CRPA) and Acinetobacter baumannii (CRAB). They can cause extremely 'difficult-to-treat' infections, while concomitantly give rise to outbreaks following dissemination in hospital settings for years. Hence patients with risk factors such as contact with health care systems outside of Scandinavia are routinely submitted to MDR screening on admission to hospitals in Scania in Sweden. Resource demanding isolation measures are upheld until negative screening results are reported.

The aim of this study is to evaluate our MDR screening in terms of the clinical course of patients with positive and negative screenings results, respectively.

Primary objective: to compare patients with positive screening results and patients with negative screening results regarding

1. admission rate within a year of screening;
2. occurrence rate of other MDR in clinical samples at the time of screening;
3. 30-day mortality and one-year mortality.

Secondary objective:

1. To evaluate the prevalence of positive screening results;
2. To characterize the MDR species and their phenotypical and genotypical resistance mechanisms;
3. To evaluate prevalence of MDR in clinical samples and time to first occurrence of phenotypically same MDR;
4. To evaluate prevalence of MDR in clinical samples within 30 days in patients with negative screening results.

For relevant primary and secondary outcomes, risk stratifications are performed for total, species and resistance mechanisms.

Methods Study design: population based observational cohort study.

Screening samples are defined as samples collected for purpose of infection prevention and control, and sent for targeted analysis of EPE, CPE, CRPA and CRAB. Following locations are typically screened: rectum/faeces, urine and risk factors such as indwelling catheters, drainage material and wound. Clinical samples are defined as all samples sent for culturing, inherently presumed for suspected infection. Isolates in clinical samples are determined as same as in screening, if they have phenotypically identical susceptibility.

Data collection: All patients included in screening (with negative and positive results) are identified through search in database (LIMS and wwBakt) at Department of Clinical Microbiology, Scania region. Social security numbers are thereafter linked to Regional Patient Register (Informationsplattformen) to collect information on comorbidities, hospital admissions, length of stay, death, antibiotics dispensed in outpatient care in general and specialised practices two weeks prior screening and up till one year after. Antibiotics during inpatient care is also collected. No medical journals will be investigated.

Condition of investigation: patients with positive screening results with following multidrug resistant gram negative bacilli: EPE, CPE, CRPA and CRAB.

"Unexposed" group consists of patients with comparable MDR risk factors but tested negative for EPE, CPE, CRPA and CRAB in screening during study time.

ELIGIBILITY:
Inclusion Criteria:

* patients with a registered screening for MDR.
* screening performed from October 1st 2013 till December 31st 2022.

Exclusion Criteria:

* carriers of MDR in question before October 1st 2013.
* patients transferred from other regions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population of Scania region in Sweden consisting of 1.4 million inhabitants. At the time of admission to a hospital in Scania, patients with risk factors for acquisition of MDR undergo screening for MDR carriage. Screenings for MDR are carried out according to local guideline "Suspected MDR - routines for hospitalized patients" and analysed and reported from the one Department of Clinical Microbiology in Lund in Scania region.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The ratio of the probability of all-cause admission in patients who are screening positive to the probability of all-cause admission in patients who are screening negative. | within one year of screening
  relative risk (RR)
The ratio of the probability of death in patients who are screening positive to the probability of death in patients who are screening negative. | 30 days and one year of screening
  relative risk (RR)
The ratio of the probability of antibiotic use in patients who are screening positive to the probability of antibiotic use in patients who are screening negative. | within one year of screening
  relative risk

SECONDARY OUTCOMES:
prevalence of positive screening results | through study completion
  number and percent
prevalence of MDR in clinical samples | through study completion
  number and percent
time to first occurrence of phenotypically same MDR as in screening | through study completion
  days, months, years
prevalence of MDR in clinical samples in patients with negative screening results | within 30 days of screening
  number and percent

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Ljungquist, M.D PhD, Principal Investigator — Region Skane

IPD SHARING:
Plan to Share IPD: Undecided
The datasets analysed during the current study will not be publicly available due to the Swedish Data Protection Act, but will probably be available from the corresponding author on reasonable request, after approval has been given by the Swedish Data Protection Agency.